CLINICAL TRIAL: NCT00541268
Title: A DANish Randomized, Controlled, Multicenter Study to Assess the Efficacy of Implantable Cardioverter Defibrillator in Patients With Non-ischemic Systolic Heart Failure on Mortality. The DANISH Study
Brief Title: Efficacy of Implantable Cardioverter Defibrillator in Patients With Non-ischemic Systolic Heart Failure on Mortality
Acronym: DANISH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Study Group (Network)
Collaborators: Danish Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2007-005606-45
Record Dates: First submitted 2007-10-09; First posted 2007-10-10 (Estimated); Last update posted 2022-04-08 (Actual); Status verified 2019-07

CONDITIONS: Heart Failure; Dilated Cardiomyopathy; Reduced LVEF
Keywords: Heart Failure; ICD; Dilated cardiomyopathy
MeSH Terms: conditions — Heart Failure; Cardiomyopathy, Dilated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A - ICD implantation (Experimental): Heart Failure nonischemic etiology treated by optimal medical treatment and receiving a prophylactic ICD
  Interventions: Device: ICD
- B - control (Active Comparator): Heart Failure nonischemic etiology treated by optimal medical treatment
  Interventions: Other: Optimal medical treatment

INTERVENTIONS:
Device: ICD — Intracardioverter defibrillators from 2 different manufacturers
  Arms: A - ICD implantation
Other: Optimal medical treatment — ACEi or angiotensin receptor blockers Betablockers Aldosterone blockers
  Arms: B - control

SUMMARY:
Primary objective: The primary objective of this study is to determine the efficacy of ICD therapy compared with control on the endpoint of death from any cause.

Secondary objective: The secondary objectives of the study are to determine if ICD therapy reduces sudden death.

Study design: Randomized, unblinded, controlled, parallel two group trial.

Primary endpoint: Time to death from any cause.

Sample size: In total, 1000 patients with 500 receiving ICD and 500 patients constituting the control group.

Summary of Subject Eligibility Criteria: Patients with clinical heart failure, left ventricular ejection fraction (LVEF) ≤ 35%, non-ischemic etiology and NT-proBNP above 200 pg/ml. Patients in NYHA class IV will only be randomised if also fulfilling criteria for a biventricular pacemaker.

Control group: Patients receiving standard therapy for heart failure including ACE-inhibitor/Angiotensin-Receptor-Blocker and Betablocker unless not tolerated. Aldosterone antagonism is optional.

Study Duration: The study comprises a screening period of up to 2 years, followed by a treatment phase of a minimum of 36 months.

Randomisation: After fulfilling all eligibility criteria, subjects will be randomized 1:1 to receive ICD implantation or continue usual control. Randomisation will be stratified according to treatment with a biventricular pacemaker.

Treatment: After randomisation patients allocated to ICD treatment should receive this as fast as possible and preferably within 2 weeks (latest 4 weeks). The ICD will be programmed with anti-tachycardia pacing and shock therapy.

Assessments: Deaths and hospitalisations for heart failure, stroke or arrhythmias will be recorded throughout the study duration.

Statistical Considerations: Median lifetime in the control group is expected to be 5 years. A p-value of 5% (2-sided) is required for significance together with a power of at least 80%. With a relative risk reduction of 25% a sample size of 812 patients in total is required. In order to allow for cross-over a sample size of 1000 is planned.

Primary Endpoint Analysis: The principal analysis for the primary endpoint (time to death from any cause) will employ the intent-to-treat principle and use a survival analysis.

Secondary Endpoint Analysis: All time-to-event secondary endpoints will be analyzed similarly to the primary endpoint.

DETAILED DESCRIPTION:
Title: A DANish randomized, controlled, multicenter study to assess the efficacy of Implantable cardioverter defibrillator in patients with non-ischemic Systolic Heart failure on mortality.

Indication: Prevention of mortality in patients at risk of sudden death.

Primary objective: The primary objective of this study is to determine the efficacy of ICD therapy compared with control on the endpoint of death from any cause.

Secondary objective: The secondary objectives of the study are to determine if ICD therapy reduces cardiovascular death as well as sudden death.

Study design: Randomized, unblinded, controlled, parallel two group trial.

Primary endpoint: Time to death from any cause.

Sample size: In total, 1000 patients with 500 receiving ICD and 500 patients constituting the control group.

Summary of Subject Eligibility Criteria: Patients with clinical heart failure, left ventricular ejection fraction (LVEF) ≤ 35%, non-ischemic etiology and NT-proBNP above 200 pg/ml. Patients in NYHA class IV will only be randomised if also fulfilling criteria for a biventricular pacemaker.

Control group: Patients receiving standard therapy for heart failure including ACE-inhibitor/Angiotensin-Receptor-Blocker and Betablocker unless not tolerated. Aldosterone antagonism is optional.

Study Duration: The study comprises a screening period of up to 2 years, followed by a treatment phase of a minimum of 36 months.

Screening and Randomisation: After the signing of informed consent, screening will include medical history, vital signs, physical exam, blood chemistry, haematology, and NT-proBNP. After fulfilling all eligibility criteria, subjects will be randomized 1:1 to receive ICD implantation or continue usual control. Randomisation will be stratified according to treatment with a biventricular pacemaker.

Treatment: After randomisation patients allocated to ICD treatment should receive this as fast as possible and preferably within 2 weeks (latest 4 weeks). The ICD will be programmed with anti-tachycardia pacing and shock therapy.

Assessments: Deaths and hospitalisations for heart failure, stroke or arrhythmias will be recorded throughout the study duration. An Endpoint Classification Committee will adjudicate hospitalizations and deaths for causality.

An independent Data Monitoring Committee will periodically review mortality data throughout the study.

Statistical Considerations: Median lifetime in the control group is expected to be 5 years. A p-value of 5% (2-sided) is required for significance together with a power of at least 80%. With a relative risk reduction of 25% a sample size of 812 patients in total is required. In order to allow for cross-over a sample size of 1000 is planned.

As event rate was lower than expected the steering committee decided to prolong follow-up and increase sample size slightly to 1150 patients. Secondly, the steering comittee decided to add cardiovascular death as a secondary outcome.

Primary Endpoint Analysis: The principal analysis for the primary endpoint (time to death from any cause) will employ the intent-to-treat principle and use a survival analysis. For each treatment group, Kaplan-Meier curves will be estimated, graphically displayed, and compared using a logrank test. A covariate-adjusted analysis of the primary endpoint using a Cox proportional hazards model will be performed as a supportive analysis. The hazard ratio and its corresponding 95% confidence interval will be estimated. Subjects withdrawing from the study early (other than for withdrawal of consent) will be followed for potential development of the primary endpoint. Subjects completing the study and not experiencing the composite event will be censored.

Secondary Endpoint Analysis: All time-to-event secondary endpoints will be analyzed similarly to the primary endpoint.

Sample Size: Hazard rates have been estimated for the placebo and ICD groups using subjects from a variety of databases (including the Echos database and the publication of Definite). Assuming a 24-month enrollment period and a 36 month follow-up period (resulting in a 5-year study with a minimum treatment period of 3 years and approximately a median survival time of 60 months), a total of 812 subjects will provide a 80% power with a 2-sided significance level of 5% for detecting a reduction in hazard of 25%.

Safety Summary: The subject incidence of adverse events will be tabulated for each group. Adverse events related to ICD implantation will be summarized. During the trial inappropriate shocks will be summarized.

Data Monitoring Committee: An independent Data Monitoring Committee consisting of members with relevant expertise will be assembled prior to study commencement. This committee will periodically review safety data.

Endpoint Classification Committee: An external Endpoint Classification Committee will adjudicate death as sudden or non-sudden throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age at the time of screening.
* Documented non-ischemic HF with an LVEF ≤ 35%.
* NYHA class II-III. If patients are planned for an implantation with a biventricular pacemaker NYHA class IV patients will be accepted for the trial.
* Before any study-specific procedure, including assessments for screening, the appropriate written informed consent must be obtained (see section 12.1).
* NT-proBNP above 200 pg/ml (see appendix D).

Exclusion Criteria:

To be eligible for this study, subjects must not meet any of the following criteria:

* Uncorrected congenital heart disease or valve obstruction, obstructive cardiomyopathy, active myocarditis, constrictive pericarditis, untreated hypothyroidism or hyperthyroidism, adrenal insufficiency, active vasculitis due to collagen vascular disease.
* On the urgent waiting list for a heart transplant (UNOS category 1A or 1B, or equivalent). Patients on the non-urgent waiting list for a heart transplant (UNOS category 2 or 7, or equivalent) are eligible for inclusion in the study.
* Recipient of any major organ transplant (eg, lung, liver, heart or kidney).
* Receiving or has received cytotoxic or cytostatic chemotherapy and/or radiation therapy for treatment of a malignancy within 6 month before randomisation or clinical evidence of current malignancy, with the following exceptions: basal or squamous cell carcinoma of the skin, cervical intraepithelial neoplasia, prostate cancer (if stable localized disease, with a life expectancy of > 2.5 years in the opinion of the investigator).
* Known to be human immunodeficiency virus positive with an expected survival of less than 5 years due to HIV.
* Renal failure treated with dialysis.
* Recent (within 3 months) history of alcohol or illicit drug abuse disorder, based on self-report
* Any condition (eg, psychiatric illness) or situation that, in the investigator's opinion, could put the subject at significant risk, confound the study results, or interfere significantly with the subject's participation in the study.
* Unwilling to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1116 (Actual)
Dates: Start 2008-02; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
All cause mortality | 5 years
  All cause mortality

SECONDARY OUTCOMES:
Cardiovascular death | 5 years
  Event committee adjudicated CV death
Sudden death | 5 years
  Event committee adjudicated sudden death
Quality of Life - Minnesota Living with Heart Failure Questionnaire | 5 years
  Patient reported outcome thru heart failure questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Lars Køber, MD, D.Sci, Study Chair — Department of Cardiology, Rigshospitalet.
Locations (4):
- Denmark (4):
  - Ålborg Sygehus, Aalborg
  - Rigshospitalet, University of Copenhagen, Copenhagen
  - Gentofte Hospital, Copenhagen
  - Odense hospital, Odense

REFERENCES:
- [Derived] Byrne C, Hasbak P, Kjaer A, Thune JJ, Kober L. Impaired myocardial perfusion is associated with increasing end-systolic- and end-diastolic volumes in patients with non-ischemic systolic heart failure: a cross-sectional study using Rubidium-82 PET/CT. BMC Cardiovasc Disord. 2019 Mar 22;19(1):68. doi: 10.1186/s12872-019-1047-x. PMID 30902043